CLINICAL TRIAL: NCT04890158
Title: Standardized Prone Positioning Compared to Usual Positioning of Very Low Birth Weight Infants Receiving Respiratory Support and the Effect on Bronchopulmonary Dysplasia
Brief Title: Prone Versus Supine Positioning and the Impact on Bronchopulmonary Dysplasia in Very Low Birth Weight Infants.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol review had expired and the study had previously been Suspended. There was no funding to continue the study.
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-13059
Record Dates: First submitted 2021-05-12; First posted 2021-05-18 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Prone Positioning; Bronchopulmonary Dysplasia
Keywords: prone positioning; bronchopulmonary dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Prone Position

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A list of study participants identified only study number, will be provided to a blinded outcomes assessor at 36 weeks post conceptional age. The respiratory support parameters of study participants will determine the primary outcome of moderate (Grade 2) or severe (Grade 3) BPD.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prone positioning for a total of 6 hours daily by study protocol (Experimental): Patients will be positioned prone for 3 hours then placed supine for 3 hours then prone again for 3 additional hours. The change in position from prone to supine and back is to more reliably document possible changes in ventilation, oxygenation, other vital signs and respiratory support required.
  Interventions: Other: Prone positioning for a total of 6 hours daily
- usual positioning (No Intervention): Patients in the newborn intensive care unit are physically handled usually every 3-4 hours. Those study participants who are randomly assigned to "usual position" may rest in a variety of positions in any order based on nursing or perceived patient preference. Positions may include supine, right lateral, left lateral, and prone as well.

INTERVENTIONS:
Other: Prone positioning for a total of 6 hours daily — Prone positioning for 6 hours daily
  Arms: Prone positioning for a total of 6 hours daily by study protocol

SUMMARY:
In this pilot study, the investigator team aims to evaluate whether standardized prone positioning compared to usual positioning improves moderate to severe bronchopulmonary dysplasia (BPD) rates as assessed at 36 weeks post conceptional age in very low birth weight preterm infants with bronchopulmonary dysplasia.

DETAILED DESCRIPTION:
The investigator team aims to enroll and randomize infants born at less than 1500 grams at birth, who remain on positive pressure support for at least 7 days after birth AND/OR on any other respiratory device such as nasal cannula with flow rates greater than 2 liters per minute (LPM) receiving supplemental oxygen of greater than 21% for at least 7 days after birth.

Patients whose families consent to participation will be assigned via block randomization to

1. usual care in which positioning and duration in each position is random per usual nursing routine OR
2. Receive standardized scheduled daily prone positioning starting on day of life 7.

As part of normal developmental care, most infants are evaluated and have care rendered (touch-time), if stable, and repositioned at set three-hour intervals to permit uninterrupted sleep and/or rest. The hands-off interval will be maintained throughout the study interval. Infants randomized to the standardized scheduled daily prone positioning will be placed in prone body position for a total of 6 hours daily, that is prone position for 3 hours, followed by supine positioning for 3 hrs, then placed in prone position for another 3-hour interval. Both infants randomized to standardized prone positioning and usual positioning will have a bedside card identifying that the infant is a study participant and will serve as a way to document the number of times any infant enrolled in the study is placed in prone positioning even if not randomized to standardized prone positioning.

Standardized daily positioning will occur for randomized patients until 36 weeks or discharge whichever is first. The primary outcome of moderate or severe BPD will be assigned by blinded study personnel based on respiratory support parameters on the day the infant is 36 weeks postconceptional age.

ELIGIBILITY:
Inclusion Criteria:

* infants born at less than 1500 grams at birth, who remain on positive pressure support for at least 7 days after birth AND/OR on any other respiratory device such as nasal cannula with flow rates greater than 2LPM receiving supplemental oxygen of greater than 21% for at least 7 days after birth. Positive pressure for the purposes of this study is defined as nasal cannula delivering a flow of 2 LPM or higher, continuous positive airway pressure (CPAP), non-invasive positive pressure ventilation or non-invasive mechanical ventilation (NIPPV/NIMV), as well infants who are intubated or have a tracheostomy for oxygenation and ventilation related to their lung disease, irrespective of the mode of ventilation.

Exclusion Criteria:

* infants who were previously on room air without a respiratory device who were intubated for the purposes of surgery and were not receiving respiratory support as defined above prior, those intubated for other airway issues such as tracheal stenosis, broncheo- or tracheomalacia, etc and not for the management of BPD. Additional patients to be excluded include those with suspected or proven genetic or other major congenital anomalies that may impact cardiac and lung function including cardiac and lung anomalies, as well as those at the time of enrollment who require surgeries that will impact their ability to be placed in prone positioning (eg gastroschisis, omphalocele, etc).

Ages: 7 Days to 14 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alecia Thompson-Branch, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prone Positioning for a Total of 6 Hours Daily by Study Protocol | Usual Positioning
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only 1 infant was enrolled (gestational age ~27 weeks), into the Prone Positioning Arm, due to early termination of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Prone Positioning for a Total of 6 Hours Daily by Study Protocol | Usual Positioning | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Customized [Count of Participants; unit: Participants]
  Approximately 27 weeks | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Moderate (Grade 2) or Severe (Grade 3) Bronchopulmonary Dysplasia
Description: The number of infants with either Moderate or Severe Bronchopulmonary Dysplasia (BPD) will be determined per study arm. Moderate and Severe BPD will be defined as follows:
  Moderate (Grade 2) BPD: If an infant requires nCPAP, NIPPV, HFNC, or NC > 2 liters per minute flow and receiving > 21% FiO2.
  Severe (Grade 3) BPD: If an infant requires invasive positive pressure ventilation via an endotracheal or tracheostomy irrespective of the amount of FiO2.
Time Frame: as determined by respiratory support requirements at 36 weeks postconceptional age
Population: The study was terminated early and Primary Outcome Measure data was not collected and/or analyzed for this study.
Arm/Group | Prone Positioning for a Total of 6 Hours Daily by Study Protocol | Usual Positioning
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Collected until the infant reaches 36 weeks preconceptional age or is discharged from the NICU, or is on 21% FiO2 (i.e., room air) without any respiratory interface, whichever is earlier.
Description: There was no enrollment into the 'Usual Positioning' arm of the study.
Arm/Group | Prone Positioning for a Total of 6 Hours Daily by Study Protocol | Usual Positioning
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/58/NCT04890158/Prot_SAP_000.pdf